CLINICAL TRIAL: NCT03332186
Title: A Phase 1, Open-Label, Parallel Group, Single-Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of BMS-986231 in Subjects With Varying Degrees of Renal Function
Brief Title: A Study of Experimental Medication BMS-986231 in Patients With Different Levels of Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV013-025
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Myocardial Failure; Cardiac Failure; Congestive Heart Failure; Kidney Failure; Renal Failure
MeSH Terms: conditions — Heart Failure; Renal Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Mild Renal Impairment (Experimental): Mild renal impairment defined as eGFR 60 to <90 mL/min/1.73 m^2
  Interventions: Drug: BMS-986231
- Moderate renal impairment (Experimental): Moderate renal impairment defined as eGFR 30 to <60 mL/min/1.73 m^2
  Interventions: Drug: BMS-986231
- Severe renal impairment (Experimental): Severe renal impairment defined as eGFR <30 mL/min/1.73 m^2, not requiring dialysis
  Interventions: Drug: BMS-986231
- Normal renal function (Experimental): Normal renal function defined as eGFR ≥90 mL/min/1.73 m^2
  Interventions: Drug: BMS-986231

INTERVENTIONS:
Drug: BMS-986231 — Intravenous infusion administration

SUMMARY:
The purpose of this study is to investigate experimental medication BMS-986231 in patients with different levels of kidney function.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Body weight ≥ 45 kg and ≤ 120 kg
* BMI ≥ 18 kg/m^2 and ≤ 35 kg/m^2
* Heart rate ≥ 50 bpm and < 95 bpm
* Stable renal impairment, defined as no clinically significant change in disease status, as documented by the subject's most recent eGFR assessment
* No changes in medication within 30 days prior to study drug administration

Exclusion Criteria:

* Clinically relevant abnormal medical history, abnormal findings on physical examination, vital signs, ECG, or laboratory tests
* History of chronic headaches, defined as occurring 15 days or more a month, over the previous 3 months
* History of headaches related to caffeine withdrawal
* History of migraine or cluster headaches
* Patients requiring dialysis will not be enrolled in this study

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) derived from plasma concentration | 11 days
Area under the concentration-time curve from time 0 extrapolated to infinity [AUC(0-inf)] derived from plasma concentration | 11 days
Metabolite ratio determined using AUC0-inf for metabolite/AUC0-inf [MRAUC(0-inf)] derived from plasma concentration | 11 days
Clearance (CL) derived from plasma concentration | 11 days
Renal clearance (CLR) derived from urine concentration | 11 days

SECONDARY OUTCOMES:
Number of adverse events (AE) | Up to 31 days
Number of serious adverse events (SAE) | Up to 31 days
Terminal elimination half-life (t1/2) | Up to 36 hours
Time of maximum observed plasma concentration (Tmax) | Up to 36 hours
AUC up to time t, where t is the last time point with concentrations above the lower limit of quantitation (AUCt) | Up to 36 hours
Terminal elimination phase rate constant (λz) | Up to 36 hours
Volume of distribution during terminal phase (Vz) | Up to 36 hours
Fraction of administered drug excreted into urine (Fe) | Up to 36 hours
Cumulative amount excreted from time 0 to the time of the last quantifiable sample (Aelast) | Up to 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- Local Institution, Prague, Czechia
- Poland (2):
  - Samodzielny Publiczny Secjalistyczny Szpital Zachodni im. sw. Jana Pawla II, Grodzisk Mazowiecki
  - Specjalistyczne Centrum Medyczne Panacea Poznan, Krakow

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm